CLINICAL TRIAL: NCT02900534
Title: Evaluation of a Randomised Guided Internet-based Self-help Intervention for Older Adults Who Seek Support for Coping With Prolonged Grief Symptoms After Marital Bereavement or Divorce - LIVIA
Brief Title: Internet-based Self-help After Spousal Bereavement or Divorce
Acronym: LIVIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Basec2016-00180
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Prolonged Grief Symptoms
Keywords: grief; depression; bereavement; divorce; online self-help
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based self-help (Experimental): The self-help programme consists of 10 text-based sessions and one supportive E-Mail a week. The programme employs cognitive-behavioural interventions. The theoretical background is the Dual Process Model by Stroebe and Schutt (1999).
  Interventions: Other: Internet-based self-help
- Waiting control group (No Intervention)

INTERVENTIONS:
Other: Internet-based self-help — 10 internet-based self-help sessions plus one supportive email a week with a cognitive-behavioural background
  Arms: Internet-based self-help

SUMMARY:
The purpose of this study is to evaluate the efficacy of an internet-based self-help intervention for older adults with prolonged grief symptoms after spousal bereavement or separation/divorce. The study design is a randomized trial with a waiting control condition of 12 weeks and a follow-up after 6 months. The investigators will test the following main hypotheses:

1. The intervention group shows a significant decrease in grief symptoms, psychological distress, depression symptoms and embitterment, and a significant increase in life satisfaction, as well as session related outcomes from baseline to 12 weeks post intervention assessment.
2. The effects in the intervention group are larger than the effects in the waiting control group.
3. These effects are stable from the post measure at 12 weeks to the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Marital bereavement or separation/divorce. Both events should have happened more than 6 months before participating in the study.
* Seeking support for coping with grief symptoms
* Internet access
* Mastery of the German language
* Informed Consent

Exclusion Criteria:

* Acute suicidality (BDI Suicide item > 1 or suicidal ideation in the telephone interview)
* No emergency plan: In the telephone interview, an emergency plan will be developed which specifies a health care professional, who participants can turn to in an acute crisis. If no such person or health care service can be found, individuals will be excluded from the intervention.
* Severe psychological or somatic disorders which need immediate treatment.
* Concomitant psychotherapy (participants may take part in the self-help intervention, but will not be included in the study.)
* Prescribed drugs against depression or anxiety lead to an exclusion if prescription or dosage has changed in the month prior or during the self-help intervention.
* Inability to follow the procedures of the study, e.g. due to comprehension problems

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05-06 (Actual); Study Completion 2018-05-06 (Actual)

PRIMARY OUTCOMES:
Grief symptoms | 12 weeks after the start of the intervention
  Texas Revised Inventory of Grief (German version, Znoj,2008; Faschingbauer, 1981)
Psychological distress | 12 weeks after the start of the intervention
  Brief Symptom Inventory (German version, Franke, 2000)
Grief symptoms | 6 months after the start of the intervention
  Texas Revised Inventory of Grief (German version, Znoj,2008; Faschingbauer, 1981)
Psychological distress | 6 months after the start of the intervention
  Brief Symptom Inventory (German version, Franke, 2000)

SECONDARY OUTCOMES:
Depression symptoms | 12 weeks after the start of the intervention
  Beck Depression Inventory II (German version, Hautzinger, Kühne & Keller, 2006)
Depression symptoms | 6 months after the start of the intervention
  Beck Depression Inventory II (German version, Hautzinger, Kühne & Keller, 2006)
Satisfaction with life | 12 weeks after the start of the intervention
  Satisfaction with life scale (German version, Schumacher, 2003)
Satisfaction with life | 6 months after the start of the intervention
  Satisfaction with life scale (German version, Schumacher, 2003)
Embitterment | 12 weeks after the start of the intervention
  Embitterment questionnaire (Znoj &, Schyder, 2014)
Embitterment | 6 months after the start of the intervention
  Embitterment questionnaire (Znoj &, Schyder, 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Hans J Znoj, Professor, Study Director — University of Bern, Switzerland
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brodbeck J, Berger T, Biesold N, Rockstroh F, Schmidt SJ, Znoj H. The Role of Emotion Regulation and Loss-Related Coping Self-efficacy in an Internet Intervention for Grief: Mediation Analysis. JMIR Ment Health. 2022 May 6;9(5):e27707. doi: 10.2196/27707. PMID 35522459
- [Derived] Brodbeck J, Berger T, Biesold N, Rockstroh F, Znoj HJ. Evaluation of a guided internet-based self-help intervention for older adults after spousal bereavement or separation/divorce: A randomised controlled trial. J Affect Disord. 2019 Jun 1;252:440-449. doi: 10.1016/j.jad.2019.04.008. Epub 2019 Apr 8. PMID 31003114
- [Derived] Brodbeck J, Berger T, Znoj HJ. An internet-based self-help intervention for older adults after marital bereavement, separation or divorce: study protocol for a randomized controlled trial. Trials. 2017 Jan 13;18(1):21. doi: 10.1186/s13063-016-1759-5. PMID 28086836